CLINICAL TRIAL: NCT00122954
Title: Fish Oil as an Adjunct Therapy for Depression in Multiple Sclerosis
Brief Title: Fish Oil for the Treatment of Depression in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Lynne Shinto, Lynn Shinto, ND, MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23AT002155-01 (NIH); K23AT002155-01 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis; Depression
Keywords: Fatty Acids, Omega-3; Fish Oils; Complementary Therapies
MeSH Terms: conditions — Multiple Sclerosis; Depression | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fish oil concentrate (Experimental): Fish oil concentrate
  Interventions: Drug: Fish oil concentrate
- Placebo oil (Placebo Comparator): Placebo oil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fish oil concentrate — fish oil concentrate at a daily dose of 6 grams (2.1 gram EPA and 1.5 gram DHA).
  Other Names: omega-3 fatty acids
  Arms: Fish oil concentrate
Drug: Placebo — soybean oil with 1% fish oil at a daily dose of 6 grams
  Arms: Placebo oil

SUMMARY:
This study will determine whether fish oil can reduce depression in people with multiple sclerosis (MS) who are mild to moderately depressed and are currently taking antidepressant medication.

Study hypothesis: Three months of fish oil supplementation will improve depression scores on the Montgomery-Asberg depression rating scale (MADRS) or Beck Depression Inventory (BDI) better than placebo.

DETAILED DESCRIPTION:
Depression occurs in 50% to 60% of all individuals with MS. Evidence suggests that the omega-3 fatty acids in fish oil supplements can significantly reduce depression with a low risk of side effects. Therefore, fish oil supplements may be a safe adjunctive therapy to improve the therapeutic benefits of antidepressants. This study will determine the effectiveness of fish oil supplements in reducing depression in MS patients who are taking antidepressant medication.

This study will last 3 months. Participants will be randomly assigned to receive either fish oil supplements or placebo daily for 3 months. At the end of 3 months, participants who show an improvement in their depressive symptoms will have the option to continue their treatment for an additional 3 months. Participants will do no respond to treatment will be excused from the study. All participants will remain on their antidepressants and MS medication throughout the study. Participants will have weekly study visits. At each visit, participants will be asked about their general health, and self-report scales will be used to assess depressive symptoms. Medication adherence will be monitored by pill counts and through red blood cell fatty acid analysis. Blood collection will occur at study start and at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting MS
* Diagnosis of depressive disorder
* Score between 11 and 30 on the Montgomery-Asberg Depression Rating Scale (MADRS)
* Score of 25 or greater on the Mini-Mental State Examination (MMSE)
* Currently taking antidepressant medication for at least 3 months prior to study entry

Exclusion Criteria:

* Currently taking fatty acid supplements
* Consume more than 6 oz of fish per week within 1 month prior to study entry
* Severe depression
* Suicidal thoughts
* Other psychological disorders
* Currently taking more than two types of antidepressants
* Any serious medical condition that would interfere with the study
* Worsening of MS symptoms or corticosteroid treatment within 1 month prior to study entry
* Current enrollment in another fish oil study
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nemets B, Stahl Z, Belmaker RH. Addition of omega-3 fatty acid to maintenance medication treatment for recurrent unipolar depressive disorder. Am J Psychiatry. 2002 Mar;159(3):477-9. doi: 10.1176/appi.ajp.159.3.477. PMID 11870016
- [Background] Su KP, Huang SY, Chiu CC, Shen WW. Omega-3 fatty acids in major depressive disorder. A preliminary double-blind, placebo-controlled trial. Eur Neuropsychopharmacol. 2003 Aug;13(4):267-71. doi: 10.1016/s0924-977x(03)00032-4. PMID 12888186
- [Background] Peet M, Horrobin DF. A dose-ranging study of the effects of ethyl-eicosapentaenoate in patients with ongoing depression despite apparently adequate treatment with standard drugs. Arch Gen Psychiatry. 2002 Oct;59(10):913-9. doi: 10.1001/archpsyc.59.10.913. PMID 12365878
- [Derived] Shinto L, Marracci G, Mohr DC, Bumgarner L, Murchison C, Senders A, Bourdette D. Omega-3 Fatty Acids for Depression in Multiple Sclerosis: A Randomized Pilot Study. PLoS One. 2016 Jan 22;11(1):e0147195. doi: 10.1371/journal.pone.0147195. eCollection 2016. PMID 26799942
- See also: Click here for more information about complementary and alternative medicine-related research at Oregon Health and Science University — http://www.ohsu.edu/xd/health/services/brain/getting-treatment/clinical-services/alternative-treatments/index.cfm
- See also: Click here for more information about research studies at the Multiple Sclerosis Center of Oregon — http://www.ohsu.edu/xd/health/services/brain/getting-treatment/diagnosis/multiple-sclerosis/index.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants randomized to the placebo group received capsules that contained soybean oil with 1% fish oil so that it was flavored to taste and smell similar to the fish oil capsules.
- Omega-3 Fatty Acids: Participants randomized to the omega-3 FA group received capsules in the form of fish oil concentrate (triglyceride form) at a daily dose of 6 grams (1.95 grams of EPA and 1.45 grams of DHA).
Period: Overall Study
Arm/Group | Placebo | Omega-3 Fatty Acids
Started | 18 | 21
Completed | 16 | 18
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants receiving soybean placebo with 1% fish oil at a daily dose of 6 grams.
- Fish Oil Concentrate: Participants receiving fish oil concentrate at a daily dose of 6 grams (2.1 grams EPA and 1.5 grams DHA)
- Total: Total of all reporting groups
Arm/Group | Placebo | Fish Oil Concentrate | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (10.0) | 50.7 (11.6) | 51.3 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease duration [Mean (Standard Deviation); unit: years] | 17.2 (10.0) | 16.6 (9.5) | 17 (10.42)
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The EDSS is an ordinal scale giving a measure of neurological impairment on a scale between 0 (normal) to 10 (dead). Patient with scores in the 0.5-4.0 range have mild disability and are able to walk at least 500 meters without aid or rest. Patients with scores > 7 cannot walk and have upper extremity dysfunction.
  units on a scale | 4.1 (2.4) | 3.2 (2.1) | 3.6 (2.3)
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: participants] — The MADRS is a structured interview assessment of depression, designed to be especially sensitive to changes in patients' depression symptoms after antidepressant therapy. The MADRS scale is more oriented towards psychic rather than somatic symptoms of depression. Scores between 11-30 indicate mild to moderate depression.
  participants | 19.1 (4.0) | 18.4 (5.3) | 18.75 (4.82)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — The BDI is a 21-item self-report measure of depression, and is commonly used in MS studies. It is an easily administered measure for depression that is not clinician-depression. Scores range from 0-63 with a higher score indicating greater depression. A score > 19 indicates moderate to severe depression.
  units on a scale | 19.6 (5.7) | 20.1 (8.0) | 19.97 (7.05)
Eicosapentaenoic Acid [Mean (Standard Deviation); unit: % total fatty acids] | 0.61 (0.3) | 0.58 (0.2) | 0.59 (0.24)
Docosahexaenoic Acid [Mean (Standard Deviation); unit: % total fatty acids] | 3.9 (1.2) | 4.0 (1.0) | 4.0 (1.0)
Adequate antidepressant use [Count of Participants; unit: Participants] — Per protocol, all participants were on one antidepressant medication. Adequate antidepressant dose is defined as minimal clinical dose to two times minimal clinical dose.
  Participants | 12 | 16 | 28
Multiple sclerosis modifying therapy (MS DMT) use [Count of Participants; unit: Participants] — MS DMT use includes: glatiramer acetate, interferon beta-1a, interferon beta-1b
  Participants | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Higher MADRS scores indicate more severe depression, and the overall score ranges from 0-60. A score of 0-6 indicates symptoms absent, 7-19 indicates mild depression, 20-34 moderate, and > 34 severe. Our primary outcome was 50% or greater improvement on the Montgomery-Asberg Depression Rating Scale (MADRS).
Time Frame: baseline to 3 months
Population: A total of 8 participants discontinued intervention (placebo n = 2, 1 colitis and 1 swallowing problems; treatment n = 6, 2 lost to follow-up, 1 bronchitis, 1 knee surgery, 1 went off antidepressant, 1 travel issues) and did not complete outcome measures
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Omega-3 Fatty Acids
Number analyzed (Participants) | 16 | 15
percentage of subjects | 45.5 | 47.4

2. Secondary Outcome: Quality of Life (SF-36)
Description: SF-36 is a commonly used measure of health-related quality of life and is well validated in many disease conditions. Responses are self-administered and responses are summed into two subscores, the mental component summary (MCS) and physical component summary (PCS). The SF-36 has eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed on a 0-100 scale. Higher scores represent higher function.
Time Frame: baseline to 3 months
Population: A total of 8 participants discontinued (placebo n = 2, 1 colitis, 1 swallowing problems; treatment n = 8, 2 lost to follow-up, 1 bronchitis, 1 knee surgery, 1 went off anti-depressant, 1 travel difficulties) and did not complete measures at end of study
Measure: Mean (Standard Error); unit: mean change of units on a scale
Arm/Group | Placebo | Omega-3 Fatty Acids
Number analyzed (Participants) | 16 | 15
mean change of units on a scale
  Physical (PCS) | -0.8 (0.8) | 1.6 (0.8)
  Mental (MCS) | 4.2 (1.0) | 1.5 (1.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to end of study at 3 months
Description: Participants were monitored twice a month (either in clinic or by phone) for general health events, worsening of depression (>30 Beck's Depression Inventory), and suicidal ideation. Worsening of depression or MS-related symptoms would result in referrals for care and withdrawal from the study. General adverse events were assessed by type, severity, relationship to supplement, action taken, and outcome.
Arm/Group | Placebo | Omega-3 Fatty Acids
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 16/18 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | Omega-3 Fatty Acids (N=21)
Urinary Tract Infection (Renal and urinary disorders) | 4 (4) | 0 (0)
multiple sclerosis relapse (Immune system disorders) | 3 (3) | 0 (0) — subject report of multiple sclerosis relapse
cold or flu (Infections and infestations) | 3 (3) | 3 (3)
bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (Immune system disorders) | 3 (3) | 0 (0) — subject reported as MS-related fatigue
numbness and tingling (Nervous system disorders) | 2 (2) | 0 (0) — MS related
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 1 (1)
arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
prolonged menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No